CLINICAL TRIAL: NCT06451900
Title: Prophylactic Role of Fenofibrate in Neonatal Jaundice
Brief Title: Role of Fenofibrate in Neonatal Jaundice
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Ibrahim, Assistant Professor of Paediatrics, Ain Shams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: prophylactic fenofibrate
Record Dates: First submitted 2024-03-11; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Neonatal Jaundice
Keywords: neonatal jaundice; prophylaxis; fenofibrate
MeSH Terms: conditions — Jaundice, Neonatal | interventions — Fenofibrate; Hypolipidemic Agents

STUDY DESIGN:
Intervention Model Description: full-term (37 to 41 weeks),Appropriate for gestational age weight between 2500 to 3500 gm infants with neonatal hyperbilirubinemia not reaching thel evel of phototherapy.The participants in our study will be divided in to three groups: Group A: full term neonates received a single oral dose of 10 mg/kg of non- micronized fenofibrate Group B: full term neonates received two oral doses of 10 mg/kg of non - micronized fenofibrate.
  Group C: full term neonates received equivalent amount of distilled water.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- fenofibrate single dose (Experimental): full term neonates will receive a single oral dose of 10 mg/kg of non- micronized fenofibrate
  Interventions: Drug: Fenofibrate
- fenofibrate double dose (Experimental): full term neonates will receive two oral doses of 10 mg/kg of non - micronized fenofibrate.
  Interventions: Drug: Fenofibrate
- placebo (Placebo Comparator): full term neonates will receive equivalent amount of distilled water.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Fenofibrate — full-term (37 to 41 weeks), Appropriate for gestational age weight between 2500 to 3500 gm infants and with neonatal hyperbilirubinemia not reaching the level of phototherapy were randomised to receive the drug in different doses or in the control group
  Other Names: lipid lowering drug
  Arms: fenofibrate double dose; fenofibrate single dose
Other: placebo — ull-term (37 to 41 weeks), Appropriate for gestational age weight between 2500 to 3500 gm infants and with neonatal hyperbilirubinemia not reaching the level of phototherapy were randomised to receive the drug in different doses or in the control group
  Other Names: control
  Arms: placebo

SUMMARY:
Fenofibrate appears to be an effective and safe drug for the treatment of neonatal hyperbilirubinemia. It has been proven that it decreases the duration of phototherapy and thus shortens the length of hospital stay.

This study was performed to study the prophylactic role of fenofibrate in prevention of neonatal jaundice.

DETAILED DESCRIPTION:
Neonatal jaundice is a common disease in neonates. Based on current statistics, 60% of term neonates and 80% of preterm neonates suffer from jaundice during the first week of birth The normal bilirubin level of the umbilical cord is 1-3 mg/dL, which increases to 5-6 mg/dL on the second to fourth days after birth and decreases to less than 2 mg/dL on the 5th to 7th days after birth .

Destruction of red blood cell and its hemoglobin component produces bilirubin which is then conjugated to a soluble form and excreted. In neonates, this becomes more significant because of high red cell mass and relative immaturity for bilirubin conjugation.

Free bilirubin deposits in the skin and mucous membranes and produces jaundice. It may also deposit in the brain where it has been implicated in causing transient dysfunction and, occasionally, permanent neuronal damage.

Every year, a huge hospital cost is imposed on parents for the treatment of neonatal jaundice. Moreover, it leads to the mother-child separation and subsequent mental health problems. Proven treatments for jaundice include phototherapy and blood exchange transfusion in which each one has its own complications . medication has also been used to prevent and treat neonatal jaundice Including IVIG, protoporphyrin, phenobarbital and fenofibrate.

Fibrates have been used for several years as a hypolipidemic drug in adults.They exert their hypolipidemic activity through peroxisome proliferator- activated receptor activation The value of this mechanism in the reduction of bile acid synthesis had been demonstrated by experimental study of cindrouk and colleagues . Fibrates also increase bilirubin conjugation and excretion via induction of glucuronyl transferase activity. Its potency to induce bilirubin conjugation is very high. Fibrates are aclass of phenoxy iso butyric acid derivatives including clofibrate and fenofibrate. Fenofibrate is one of the fibrates it has inducing effect on glucuronyl transferase activity, it increases bilirubin conjugation and excretion making it possible to be used in the treatment of neonatal jaundice via influencing bilirubin metabolism. Fenofibrate is very similar to clofibrate in its action. However, it is simply more accessible and has more safety profile, therefore, it is much safer to be given to children than clofibrate. Fenofibrate has been used in treatment of neonatal jaundice the researchers aim to explore its efficiency as a prophylactic agent in neonates with neonatal jaundice not reaching the level of phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* full-term (37 to 41 weeks),
* Appropriate for gestational age weight between 2500 to 3500 gm infants
* neonatal hyperbilirubinemia not reaching the level of phototherapy.

Exclusion Criteria:

* Newborns with congenital malformations.
* Conjugated hyperbilirubinemia.
* Newborns who need exchange transfusion and phototherapy.
* Newborns presenting with ABO or Rh incompatibility.
* G6PD deficiency.
* Newborns with skin abrasions or infections.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
change in total serum bilirubin | up to 5 days
  Decline in total serum bilirubin values per unit of time after 12, 24, 36, 48 hours, 5 days from intervention.
start of phototherapy | up to 5 days
  time at which phototherapy will be initiated from receiving the drug and till 5 days later
start of exchange transfusion | up to 5 days
  time at which patient needed to perform exchange transfusion after receiving the drug till five days later

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No
data will be provided when requested appropriately for reasonable reasons from the main investigator